CLINICAL TRIAL: NCT06881264
Title: A Randomized, Open-label, Parallel, Treat to Target Study Comparing the Efficacy and Safety of HR17031 With Insulin Glargine in Chines Subjects With Type 2 Diabetes Inadequately Controlled With Metformin in Combination With or Without Another Oral Antidiabetic Drug (OAD)
Brief Title: A Study Comparing HR17031 With Insulin Glargine in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR17031-301
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Adult Patients With Type 2 Diabetes Uncontrolled on Oral Antidiabetic Drugs
MeSH Terms: interventions — Insulin Glargine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: HR17031 injection (Experimental)
  Interventions: Drug: HR17031 injection
- Treatment group B: insulin glargine (Experimental)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: HR17031 injection — HR17031 injection
  Arms: Treatment group A: HR17031 injection
Drug: insulin glargine — insulin glargine
  Arms: Treatment group B: insulin glargine

SUMMARY:
The aim of this trial is to confirm the efficacy of HR17031 in controlling glycaemia in Chinese subjects with type 2 diabetes mellitus inadequately controlled on oral antidiabetic agents

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-75 years at the time of signing the informed consent (both ends included);
2. Body Mass index (BMI) of 20.0-40.0 kg/m2 (both ends included);
3. Diagnosed with type 2 diabetes for at least 90 days prior to screening;
4. Tested by local laboratory, HbA1c is 7.5%-11% (including both ends);
5. Before screening, the daily basal insulin dose had been stabilized at 20-40 U/day (including both ends) for at least 60 days;
6. When screening: ① metformin monotherapy stable treatment ≥ 3 months; or ② metformin combined with another OAD for stable treatment for ≥ 3 months; Metformin dose ≥ 1500 mg/day or maximum tolerated dose.
7. Ability and willingness to comply with protocol requirements, including self-monitoring of blood glucose, recording subject diary, and using pre-filled injection pen.

Exclusion Criteria:

1. Known or suspected allergy to the investigational drug product or its components or excipients;
2. Systemic glucocorticoid use within 3 months prior to screening;
3. Use of weight loss drugs within 3 months prior to screening;
4. Received insulin therapy within 1 year prior to screening (excluding short-term therapy [continuous treatment ≤14 days] or insulin therapy for gestational diabetes);
5. Cardiovascular disease, defined as congestive heart failure (NYHA III-IV), unstable angina pectoris, stroke (except lacunar infarction without symptoms), myocardial infarction, coronary revascularization within 6 months prior to screening; And/or coronary, carotid, or peripheral arterial revascularization is planned at screening;
6. (with or without treatment) uncontrolled severe hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg);
7. Proliferative retinopathy or macular degeneration requiring acute treatment, painful diabetic neuropathy, diabetic foot ulcers, intermittent claudication at screening;
8. Patients diagnosed with mental disorders; Mentally incapacitated or speech impediment, unable to fully understand the trial protocol or unwilling to collaborate;
9. Known or suspected abuse of alcohol or narcotics;
10. Previous history of pancreatitis (acute or chronic);
11. During pregnancy or lactation;fertile women (WOCBP) or men who have fertility plan or unwilling to use appropriate contraceptive methods from the signing of the informed consent to 3 months after last use of the investigational drug product;
12. Any condition, determined by the investigator, interfere with the efficacy or safety results of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c: Changes in HbA1c from baseline to week 26 | week 26

SECONDARY OUTCOMES:
Proportion of subjects achieved HbA1c<7.0% at week 26 | at week 26
Change in body weight from baseline after 26 weeks of treatment | 26 weeks
Proportion of subjects achieved HbA1c<7.0% without body weight gain at week 26 | week 26
Actual Daily Insulin dose at week 26 | week 26
Proportion of subjects achieved HbA1c≤6.5% at week 26 | week 26
Changes in Fasting Plasma Glucose (FPG) after 26 weeks of treatment | 26 weeks
Proportion of subjects achieved HbA1c≤6.5%without body weight gain at week 26 | week 26
Proportion of subjects achieved HbA1c<7.0% without Level 2 and Level 3 hypoglycemic event after 12weeks treatment | 12weeks
Proportion of subjects achieved HbA1c≤6.5% without Level 2 and Level 3 hypoglycemic event after 12weeks treatment | 12weeks
Proportion of subjects achieved HbA1c<7.0% without body weight gain and without Level 2 and Level 3 hypoglycemic event after 12weeks treatment at week 26 | at week 26
Proportion of subjects achieved HbA1c≤6.5% without body weight gain and without Level 2 and Level 3 hypoglycemic event after 12weeks treatment at week 26 | at week 26
Proportion of subjects achieved HbA1c<5.7% at week 26 | at week 26
Change in mean of the 7-point SMPG profile from baseline (week 0) to week 26; | week 26;
Change from baseline (week 0) in post-prandial SMPG increments for all meals after 26 weeks of treatment | 26 weeks
Changes in HbA1c from baseline after 52 weeks of treatment | 52 weeks
Changes in FBG from baseline after 52 weeks of treatment | 52 weeks
Changes in body weight from baseline after 52 weeks of treatment | 52 weeks
Proportion of subjects achieved HbA1c<7% at week 52 | at week 52
Proportion of subjects achieved HbA1c≤6.5% at week 52 | at week 52
Proportion of subjects achieved HbA1c<7% without body weight gain at week 52 | at week 52
Proportion of subjects achieved HbA1c≤6.5% without body weight gain at week 52 | at week 52
Proportion of subjects achieved HbA1c<7.0% without Level 2 and Level 3 hypoglycemic event after 12weeks treatment at week 52 | at week 52
Proportion of subjects achieved HbA1c<7.0% without body weight gain and without Level 2 and Level 3 hypoglycemic event after 12weeks treatment at week 52 | at week 52
Proportion of subjects achieved HbA1c≤6.5% without body weight gain and without Level 2 and Level 3 hypoglycemic event after 12weeks treatment at week 52 | at week 52
Proportion of subjects achieved HbA1c<5.7% at week 52 | at week 52
Change in mean of the 7-point SMPG profile from baseline (week 0) to week 52 | week 52
Change from baseline (week 0) in post-prandial SMPG increments for all meals after 52 weeks of treatment | 52 weeks
Actual Daily Insulin dose at week 52 | at week 52
Number of Treatment-emergent Hypoglycemic event from screening to week 53 | from screening to week 53
Number of Treatment-emergent Adverse Events from screening to week 53 | from screening to week 53
Number of participants who were assessed for anti-insulin glargine antibodies, anti-INS068 antibodies and anti-HR20004 antibodies at week 27 | at week 27

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided